CLINICAL TRIAL: NCT00727753
Title: Effects of Vascular Endothelial Growth Factor Antagonism With Ranibizumab or Bevacizumab in Patients With Neovascular Macular Degeneration
Brief Title: VEGF-antagonism and Endothelial Function in Age-related Macular Degeneration (AMD)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-770
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; Age-Related Maculopathies
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ranibizumab
  Interventions: Drug: Ranibizumab
- Bevacizumab
  Interventions: Drug: Bevacizumab
- Dry AMD
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Ranibizumab — ranibizumab (0.5 mg) will be injected intraocular
  Other Names: Lucentis
  Groups: Ranibizumab
Drug: Bevacizumab — Bevacizumab (1.25 mg) will be injected intraocular
  Other Names: Avastin
  Groups: Bevacizumab
Other: No treatment — No treatment
  Groups: Dry AMD

SUMMARY:
The objective of this study is to evaluate the effects of 2 intravitreal injections with Ranibizumab or Avastin on endothelial function in subjects with neovascular macular degeneration compared to patients with dry AMD.

ELIGIBILITY:
Inclusion Criteria for active treatment:

* Age: 50 - 80 years
* Diagnosis of neovascular macular degeneration suitable for intravitreal anti-VEGF therapy
* Stable medication for general conditions for at least 1 month
* Written informed consent for participation in the study

Inclusion criteria for controls:

* Age: 50 - 80 years
* Diagnosis of "dry" AMD
* "dry" AMD is defined as at least Age-Related-Eye-Disease-Study (AREDS) category 2 in both eyes and no evidence of neovascularization in either eye
* Stable medication for general conditions for at least 1 month
* Written informed consent for participation in the study

Exclusion Criteria for all subjects:

* Myocardial infarction, unstable angina, stroke within 3 months prior to study entry
* Thoracic or cardiac surgery and/or coronary intervention/revascularisation procedure (within 3 months before randomization)
* Uncontrolled symptomatic congestive heart failure (NHYA> II) in the last 4 weeks prior to study
* Renal insufficiency (Creatinine Clearance < 50ml/min)
* Ventricular tachyarrhythmias
* Poorly controlled hypertension, defined as resting blood pressure ≥ 160/100 mmHg
* Symptomatic hypotension
* Long acting nitrates
* Smoking (>5 Zig./d)
* Diabetes mellitus
* Dyslipidemia (LDL-cholesterol > 4.5 mmol/l)
* Liver disease (ALT or AST >3x ULN)
* Alcohol or drug abuse
* Hypersensitivity to the active substance or to any of the excipients
* Active or suspected ocular or periocular infections
* Patients with active severe intraocular inflammation
* Malignancy (unless healed or remission > 5 years)
* Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
* Participation in another study within the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See eleigibility criteria
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change of endothelial function after 2 intravitreal injections and 8 weeks follow-up with ranibizumab or bevacizumab in patients with neovascular macular degeneration compared to patients with dry AMD. | 8 weeks

SECONDARY OUTCOMES:
Change in cardiovascular and ophthalmological parameters. | 8 weeks
  Secondary outcomes include evaluation of retinal thickness as measured by optical coherence tomography (OCT), change in best-corrected visual acuity (BCVA), "Early Treatment Diabetic Retinopathy Study" (ETDRS) letters, ambulatory blood pressure, vascular compliance, biomarkers of vascular function and platelet function.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, Prof MD, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland